CLINICAL TRIAL: NCT06491511
Title: Non-Invasive Transcutaneous Repetitive Phrenic Nerve Stimulation Assessment in Critically Ill Patients Under Mechanical Ventilation - Pilot Study
Brief Title: Repetitive Phrenic Nerve Stimulation in Critically Ill Patients Under Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Sung Eun Hyun, Assistant professor (MD, PhD), Seoul National University Hospital
Other Study IDs: 2312-166-1498
Record Dates: First submitted 2024-06-14; First posted 2024-07-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Phrenic Nerve; Electrical Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ICU patients: ICU patient with mechanical ventilator
  Interventions: Procedure: Transcutaneous, repetitive phrenic nerve electrical stimulation

INTERVENTIONS:
Procedure: Transcutaneous, repetitive phrenic nerve electrical stimulation — Phrenic nerve electrical stimulation with different stimulation intensity and frequency

SUMMARY:
Subjects: Patients aged 19 and older who are currently in the ICU and undergoing invasive mechanical ventilation.

Methods: The study involves performing non-invasive repetitive phrenic nerve stimulation in ICU patients on mechanical ventilation.

Stimulation protocol: The intensity and position of phrenic nerve stimulation were individualized. The frequency was set to 10Hz, 15Hz, and 20Hz. The duration of stimulation was adjusted according to the set inspiration time of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 and older who are admitted to the ICU at Seoul National University Hospital
* Patients receiving invasive mechanical ventilation (via endotracheal tube or tracheostomy)
* Patients who have been on invasive mechanical ventilation (via endotracheal tube or tracheostomy) for more than 48 hours
* Patients who have listened to and understood the explanation of the purpose and procedures of the study and have voluntarily agreed to participate. In cases where the patient has impaired consciousness or cognitive function and is unable to consent, the patient's legal representative has agreed to the patient's participation in the study.

Exclusion Criteria:

* Patients with implanted or externally applied electrical devices (such as pacemakers, defibrillators, implantable defibrillators, vagus nerve stimulators, spinal cord stimulators, gastric stimulators, diaphragm stimulators, etc.)
* Patients with a history of neck tumors, cervical spine instability, or neck surgery
* Patients with internal jugular vein catheters, infections, or inflammatory signs at the electrical stimulation site, making percutaneous phrenic nerve access impossible
* Patients with neurological or neuromuscular diseases that significantly affect respiratory muscle function
* Patients currently receiving neuromuscular blocking agents
* Patients already diagnosed with or suspected of having phrenic nerve paralysis
* Patients with elevated hemidiaphragm observed on chest X-ray
* Patients with pleural effusion occupying more than one-third of the pleural space or pneumothorax requiring chest tube insertion, as seen on chest X-ray
* Patients who are confirmed or presumed to be pregnant
* Patients with a body mass index (BMI) ≥ 40
* Patients for whom life-sustaining treatment has been decided to be withdrawn and who have no plans for active treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patients aged 19 and older who are admitted to the ICU at Seoul National University Hospital on invasive mechanical ventilation for more than 48 hours
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Maximum diaphragm thickness during phrenic nerve repetitive stimulation | Measured one time between 48 hours after intubation and before extubation.
  Maximum diaphragm thickness (mm)
Change in diaphragm thickness before and during phrenic nerve repetitive stimulation | Measured one time between 48 hours after intubation and before extubation.
  Change of diaphragm thickness (mm)

SECONDARY OUTCOMES:
Amplitude of the phrenic nerve compound motor action potential during phrenic nerve repetitive stimulation | Measured one time between 48 hours after intubation and before extubation.
  CMAP amplitude (mV)
Area of the phrenic nerve compound motor action potential during phrenic nerve repetitive stimulation | Measured one time between 48 hours after intubation and before extubation.
  CMAP area (ms*mV)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Eun Hyun, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided